CLINICAL TRIAL: NCT05796180
Title: The Effect of Sexual Health Counseling Based on the BETTER Model on Postpartum Sexual Life Quality: A Randomized Controlled Study
Brief Title: Sexual Health Counseling Based on the BETTER Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Nurgül ŞİMAL YAVUZ, Lecturer, Lokman Hekim University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: NSIMALYAVUZ
Record Dates: First submitted 2023-02-22; First posted 2023-04-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Health Knowledge, Attitudes, Practice; Sexuality
Keywords: Sexual Health Counseling; Sexual Life Quality; Postpartum; Postpartum Sexual Life Quality; BETTER Model
MeSH Terms: conditions — Behavior; Sexuality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral: sexual health counseling based on the BETTER model (Experimental): Sexual health counseling based on the BETTER model
  The content of the research will be discussed by face-to-face interviews with women who gave birth vaginally and applied to the hospital for birth control 8-10 weeks after delivery. Pre-evaluation forms will be applied to women who have agreed to participate in the study to evaluate the inclusion criteria. Women who meet the inclusion criteria will be divided into experimental-control groups using the block randomization method.
  An appointment will be made for interviews with the women in the experimental group. It is planned that these meetings will be held in the form of online video calls and will last an average of 45 minutes. The final tests will be held 8 weeks after the online meetings are over.
  Interventions: Behavioral: Behavioral: sexual health counseling based on the BETTER model
- Control group: Routine postpartum care (No Intervention): Routine postpartum care
  Women who gave birth vaginally and applied to the hospital for postpartum controls 8-10 weeks after delivery will be interviewed face-to-face with the women and the content of the research will be mentioned. Pre-evaluation forms will be applied to the women who accepted to participate in the study to evaluate the inclusion criteria. Women who meet the inclusion criteria will be divided into experimental-control groups using the block randomization method. Women in the control group will receive routine postpartum care administered in the hospital. Women in the control group will receive routine postpartum care administered in the hospital. Post-tests will be administered 8 weeks after the first interview.

INTERVENTIONS:
Behavioral: Behavioral: sexual health counseling based on the BETTER model — The content of the research will be discussed by face-to-face interviews with women who gave birth vaginally and applied to the hospital for birth control 8-10 weeks after delivery. Pre-evaluation forms will be applied to women who have agreed to participate in the study to evaluate the inclusion criteria. Women who meet the inclusion criteria will be divided into experimental-control groups using the block randomization method.
  An appointment will be made for interviews with the women in the experimental group. It is planned that these meetings will be held in the form of online video calls and will last an average of 45 minutes. The final tests will be held 8 weeks after the online meetings are over.
  Arms: Behavioral: sexual health counseling based on the BETTER model

SUMMARY:
In this study, the investigators wanted to examine the effect of sexual health counseling to women in the postpartum period on the quality of life of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous,
* Weeks of gestation 37 weeks and over,
* Who had a singleton pregnancy,
* Having a sexual partner/partner,
* Having started sexual intercourse before starting training,
* Without a diagnosed chronic disease (DM, HT, Heart disease, etc.),
* Labour week 37 weeks and over
* 18 years or older,
* Able to speak and understand Turkish,

Exclusion Criteria:

* Edinburgh Postpartum Depression Scale score of 12 and above,
* To have received training on sexual health and family planning in a hospital or other health institution other than discharge training,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-02-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Postpartum Sexual Life Quality Scale | 8 week
  The scale is still under development.
Arizona Sexual Experiences Scale | 8 week
  The Arizona Sexual Experiences Scale (ASEX) is a 6-point Likert-type self-report scale and consists of 5 questions. This form reveals the capacity to reach orgasm, the feeling of satisfaction, vaginal wetness, arousal and sexual drive. Each question is scored from 1 to 6. The total score ranges from 5 to 30. Low scores indicate that the sexual response is satisfactory, strong and easy, while high scores indicate the presence of sexual dysfunction. The total scale score is formed by the sum of the scores of the scale items in the scale. The cut-off point of the scale was determined as 11. A score of 5 or more for each item indicates that there is a sexual dysfunction related to that item.
VAS satisfaction scale | 8 week
  Women's satisfaction with sexual life will be evaluated with the visual analog scale (VAS). It shows that women who score high on the scale, which is scored between 0 (very dissatisfied) and 10 (very satisfied), also have high sexual satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Nurgül ŞİMAL YAVUZ, Lecturer, Study Director — Lokman Hekim University
Locations (1):
- Lokman Hekim Etlik Hospital, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No